CLINICAL TRIAL: NCT02692378
Title: A Feasibility Randomised Controlled Trial: Effects of Oral Sodium Bicarbonate Supplementation in Patients on Haemodialysis
Brief Title: Effects of Oral Sodium Bicarbonate Supplementation in Haemodialysis Patients (BicHD)
Acronym: BicHD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Imperial College Healthcare NHS Trust (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 15HH2613
Record Dates: First submitted 2016-02-23; First posted 2016-02-26 (Estimated); Last update posted 2016-10-03 (Estimated); Status verified 2015-11

CONDITIONS: End-stage Renal Disease
Keywords: Haemodialysis; sodium bicarbonate; potassium; arrhythmia; muscle; symptoms
MeSH Terms: conditions — Kidney Failure, Chronic; Arrhythmias, Cardiac | interventions — Sodium Bicarbonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment (Active Comparator): Standard haemodialysis treatment thrice weekly (using a standard dialysate containing bicarbonate at a concentration of 35mmols/L) with the addition of oral sodium bicarbonate 500mg capsules for 12 weeks (weeks 5-16 of the study).
  The dosage will be titrated to individual blood levels. Starting dose will be 1g twice daily and if predialysis bicarbonate levels remain <22mmols/L the dose will be increased by 0.5g twice daily each week. The maximum dose would be 3g twice daily.
  The oral sodium bicarbonate may be withheld on dialysis days, when bicarbonate will be supplemented through the dialysate. This will be assessed on a case by case basis.
  Interventions: Drug: sodium bicarbonate 500mg capsules
- Control (No Intervention): Standard haemodialysis treatment thrice weekly using a standard dialysate containing bicarbonate at a concentration of 35mmols/L.

INTERVENTIONS:
Drug: sodium bicarbonate 500mg capsules — Defined by active substance and brand names not specified in protocol
  Arms: Treatment

SUMMARY:
The purpose of the study is to investigate whether oral sodium bicarbonate supplementation to ensure a constant bicarbonate profile in haemodialysis patients will primarily lower predialysis potassium levels and secondary lead to improvements in cardiac function, muscle mass and dialysis related symptoms.

DETAILED DESCRIPTION:
Background:

One of the functions of dialysis is to correct electrolyte abnormalities which occur with renal failure, such as variations in potassium and bicarbonate levels, which are linked to important clinical outcomes for patients. Metabolic acidosis, reflected by falling bicarbonate levels, is a frequent event in haemodialysis patients and its correction is one of the goals of effective dialysis. Bicarbonate replacement is routinely delivered during each dialysis session thrice weekly with the use of high dialysate bicarbonate. However, local and national data show that over 50% of patients fail to meet a bicarbonate level within the normal range before each dialysis session. Low predialysis bicarbonate levels of less than 22mmols/L have been linked with increased all-cause mortality in haemodialysis patients.

Evidence from previous studies suggests that a continuous replacement (i.e. daily) with oral sodium bicarbonate capsules may be a superior correction of acidosis to the current treatment of intermittent replacement during dialysis.

Aims and objectives:

This randomised controlled study aims to investigate the effects of oral sodium bicarbonate supplementation on:

Primary objective: Pre and post dialysis potassium without increasing intradialytic potassium gradient.

Secondary objectives:

1. Risk of arrhythmia as measured by ECG analysis
2. Muscle mass as measured by body composition monitoring
3. Muscle function as measured by handgrip strength
4. Haemodialysis related cramps as measured by a symptom scale-renal questionnaire

Patients will be recruited from Imperial College Healthcare NHS (National Heath Service) Trust haemodialysis units and randomised to two equally numbered groups. One group will receive the standard dialysis treatment (control) and the other one will receive the standard dialysis with the addition of capsules of sodium bicarbonate (intervention). The dose of sodium bicarbonate will be adjusted according to individual levels. The study duration is 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

Patients on haemodialysis for at least 3 months, Patients who primarily have predialysis bicarbonate levels of less than 22mmols/L over the last 6 months, Patients who are not already taking oral sodium bicarbonate, Able and willing to provide written informed consent

Exclusion Criteria:

Patients who primarily have predialysis potassium levels of less than 4mmols/L over the last 6 months, Patients who are already taking oral sodium bicarbonate, Patients on lithium, Bedbound patients, Pregnant patients, Dementia, Recurrent hospital admissions, Non-English speaking and unable to provide written informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2015-11; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
pre dialysis potassium level and intradialytic potassium gradient | 12 weekly blood tests over a period of 16 weeks
  Measurements over the first 4 weeks to establish blood potassium profile. Measurements over weeks 5-8 to detect early blood changes. Measurement over weeks 13-16 to detect late blood changes.

SECONDARY OUTCOMES:
12 lead Electrocardiogram analysis | 3 timepoints (weeks 4, 8 and 16) over a period of 16 weeks
  Electrocardiogram analysis before and after dialysis for the measurement of QT dispersion. Increase of the QT dispersion is linked to risk of ventricular arrhythmias.
Total body muscle mass | 2 timepoints (weeks 4 and 16) over a period of 16 weeks
  Body composition measurement before dialysis with the validated body composition monitor by Fresenius
Handgrip strength | 2 timepoints (weeks 4 and 16) over a period of 16 weeks
  Handgrip strength to measure muscle function. Measured before dialysis with the ®Jamar handgrip dynamometer.
Symptom severity | 3 timepoints (weeks 4,8 and 16) over a period of 16 weeks
  Haemodialysis related symptoms measured by a validated palliative outcome symptom scale-renal questionnaire (POS-S)

CONTACTS AND LOCATIONS:
Overall Officials: Damien Ashby, PhD, MRCP, Principal Investigator — Imperial College Healthcare NHS Trust
Locations (1):
- Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bleyer AJ, Russell GB, Satko SG. Sudden and cardiac death rates in hemodialysis patients. Kidney Int. 1999 Apr;55(4):1553-9. doi: 10.1046/j.1523-1755.1999.00391.x. PMID 10201022
- [Background] Bossola M, Giungi S, Tazza L, Luciani G. Long-term oral sodium bicarbonate supplementation does not improve serum albumin levels in hemodialysis patients. Nephron Clin Pract. 2007;106(1):c51-6. doi: 10.1159/000101484. Epub 2007 Apr 2. PMID 17409769
- [Background] Brady JP, Hasbargen JA. Correction of metabolic acidosis and its effect on albumin in chronic hemodialysis patients. Am J Kidney Dis. 1998 Jan;31(1):35-40. doi: 10.1053/ajkd.1998.v31.pm9428449.
- [Background] Brass EP, Adler S, Sietsema KE, Amato A, Esler A, Hiatt WR. Peripheral arterial disease is not associated with an increased prevalence of intradialytic cramps in patients on maintenance hemodialysis. Am J Nephrol. 2002 Sep-Dec;22(5-6):491-6. doi: 10.1159/000065285. PMID 12381949
- [Background] Cupisti A, Galetta F, Caprioli R, Morelli E, Tintori GC, Franzoni F, Lippi A, Meola M, Rindi P, Barsotti G. Potassium removal increases the QTc interval dispersion during hemodialysis. Nephron. 1999 Jun;82(2):122-6. doi: 10.1159/000045387. PMID 10364703
- [Background] Graham KA, Reaich D, Channon SM, Downie S, Goodship TH. Correction of acidosis in hemodialysis decreases whole-body protein degradation. J Am Soc Nephrol. 1997 Apr;8(4):632-7. doi: 10.1681/ASN.V84632. PMID 10495793
- [Background] Heguilen RM, Sciurano C, Bellusci AD, Fried P, Mittelman G, Rosa Diez G, Bernasconi AR. The faster potassium-lowering effect of high dialysate bicarbonate concentrations in chronic haemodialysis patients. Nephrol Dial Transplant. 2005 Mar;20(3):591-7. doi: 10.1093/ndt/gfh661. Epub 2005 Feb 1. PMID 15687112
- [Background] Ikizler TA, Pupim LB, Brouillette JR, Levenhagen DK, Farmer K, Hakim RM, Flakoll PJ. Hemodialysis stimulates muscle and whole body protein loss and alters substrate oxidation. Am J Physiol Endocrinol Metab. 2002 Jan;282(1):E107-16. doi: 10.1152/ajpendo.2002.282.1.E107. PMID 11739090
- [Background] Movilli E, Viola BF, Camerini C, Mazzola G, Cancarini GC. Correction of metabolic acidosis on serum albumin and protein catabolism in hemodialysis patients. J Ren Nutr. 2009 Mar;19(2):172-7. doi: 10.1053/j.jrn.2008.08.012. PMID 19218045
- [Background] Vashistha T, Kalantar-Zadeh K, Molnar MZ, Torlen K, Mehrotra R. Dialysis modality and correction of uremic metabolic acidosis: relationship with all-cause and cause-specific mortality. Clin J Am Soc Nephrol. 2013 Feb;8(2):254-64. doi: 10.2215/CJN.05780612. Epub 2012 Nov 26. PMID 23184567